CLINICAL TRIAL: NCT02175147
Title: Patient-centred Integrated Palliative Care Pathways in Advanced Cancer and Chronic Disease
Acronym: InSup-C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: European Union (Other); Medical University of Pecs (Other); Lancaster General Hospital (Other); University Hospital, Bonn (Other); KU Leuven (Other); World Health Organization (Other); European Association for Palliative Care (Unknown); University of Rotterdam, The Netherlands (Other); University of Navarra (Other); University of Sheffield (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: 305555
Record Dates: First submitted 2014-06-02; First posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: COPD; Cancer; Heart Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Neoplasms; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Rationale: Palliative care integration in treatment pathways, palliative care networks and institutional collaborations in health services delivery seems a promising approach reducing fragmentation and discontinuity. Integrated Palliative Care (IPC) approaches in Europe are largely unknown and under-investigated. The investigators aim is to explore experiences of patients with advanced cancer, Chronic Obstructive Pulmonary Disease (COPD) and Chronic Heart Failure (CHF), family and professional caregivers within with IPC. This includes perceived quality of life, quality of care, burden/rewards of care giving, symptoms and collaboration between caregivers in the patient's care network.

Objectives: To investigate how patients with advanced cancer, COPD and CHF, their family and professional caregivers within a selection of IPC initiatives in Belgium, Germany, Hungary, The Netherlands and United Kingdom experience care delivery in the last phase of disease.

* To investigate what opinions patients and family caregivers have on the (continuity and) quality of care delivered
* To investigate how patients rate their symptoms and quality of life
* To investigate how family caregivers rate their burden / rewards of care giving
* To investigate how the care network of the patient is organised with respect to the type, properties and quality of relationships between patients and family / professional caregivers

Study design: Longitudinal multiple embedded case study.

Study population: Adult patients with advanced cancer, COPD, and CHF under the care of IPC initiatives in five participating countries, their family and professional caregivers. The investigators aim to enroll up to 288 patients, 288 family caregivers and 192 professional caregivers in total.

Study parameters: Experiences with IPC initiatives, quality of care, quality of life, perceived symptoms, perceived collaboration between professional caregivers, burden and rewards of care giving.

Methods: Semi-structured interviews, patient diary, Social Network Analysis and the following questionnaires: Palliative care Outcome Scale; Canhelp Lite, Caregiver Reaction Assessment. Patients and family caregivers will be followed over 3 months at 4 consecutive contact points. The diary (containing two questions) will be kept weekly by patients. There will be group or individual interviews with professional caregivers.

Analysis: The overall analysis will involve a synthesis of the qualitative and quantitative data. For more information see Detailed Description.

DETAILED DESCRIPTION:
Monitoring and Quality Assurance:

Training for researchers:

In order to ensure the best quality of the study, researchers will take part in at least two compulsory training sessions. During the training ethical and professional issues will also be discussed, such as:

* ethical issues (e.g. handling vulnerable groups in interview situations)
* data management (protection of privacy of medical and research records)
* interview training in order to standardise interview techniques
* how to analyse qualitative and quantitative data, and how to synthesize them in this research (to the analysing researchers in the partner countries).

Qualitative data:

Interviews will be tape recorded and transcribed verbatim, and will be evaluated with content analysis using qualitative software package NVivo 10. After two pilot interviews responsible researchers from each partner country will discuss a preliminary code book. These codes and themes will form the basis of the coding strategy throughout data collection and the data analysis. Analysis will be ongoing throughout the fieldwork in order to allow emergent themes to be fed back into the data collection. During data collection new relevant codes will be included in the code book.

The interviews will be coded in the national languages of the five countries under examination. This will result in five country reports about the experiences of patients with advanced cancer, COPD and CHF, their family and professional caregivers within a selection of IPC initiatives in the particular country with the care delivery in the last phase of disease. These country reports will be translated into English and will be analysed and result in one overall report.

Quantitative data:

Statistical analysis will be performed using SPSS Statistics 20. The investigators will use descriptive statistics such as frequencies, crosstabs, means, standard deviation. The quantitative data will be used as a background description of the population. The overall analysis will involve a synthesis of the qualitative and quantitative data. During the analysis phase the investigators will integrate the quantitative variables, qualitative findings and evaluations in order to get complete insight in the topic.

Treatments for missing data:

The investigators will use the following approach to missing data: to omit questions with missing data and to perform analyses of questions on what remains. Missing data will be accounted for in the analysis and the implications will be made clear.

Handling and storage of data and documents:

The confidentiality of data collected within the patient study will be secured according to national and European regulation. Data from patients will be anonymised and disclosure of information from the study to third parties will be limited to those undertaking legitimate peer review of the scientific and ethical aspects of the study, co-workers and patients, so that consent can be obtained and customary medical care can be provided.

Patient confidentiality and welfare will always be maintained as the highest priority. All data gathered and documents will be stored anonymously. Each patient, family caregiver and professional caregiver will be allocated a unique identification number. No identifying information linking the person and identification number will be kept on the data base. The investigators will analyze data by identification number only. Patient data will be stored in a protected database with log function. The master database will be kept at the centre of the research coordinator of the Radboud University Medical Centre.

Assessment of progress and quality:

Researchers (who will do fieldwork at IPC initiatives involved) will report fieldwork progress (patient recruitment and data collection) and the quality of data collected every other week to their lead researcher (who is responsible for the research in the particular country). Contents of the progress and quality report:

1. Number of persons (patients and family caregivers) involved
2. Number of completed questionnaires and interviews
3. Quality of completed questionnaires and interviews
4. Attrition (death of patients, early terminated interviews)
5. Other research-related events (e.g. delays)

Lead researchers will summarize researches' reports and send a progress and quality report to the study principal investigator every month (The study principal investigator is responsible for the research in the framework of InSup-C project.)

The study principal investigator organizes a 3-monthly structure of (tele)conference to monitor progress and quality and to report this to the Project Management Office (PMO). The PMO works under supervision of the Executive Board of the project. The PMO will provide the Executive Board with project process reports at least every six months or more frequently if necessary.

Annual progress report:

The Principal Investigator will submit a summary of the progress of the study to the accredited ethical committee once a year. Information will be provided on the date of inclusion of the first subject, numbers of subjects included and numbers of subjects that have completed the trial, (serious) adverse events, other problems, and amendments.

End of study report:

The Principal Investigator will notify the accredited ethical committee of the end of the study within a period of eight weeks. The end of the study is defined as the last study participant's last interview. In case the study is ended prematurely, the responsible researcher will notify the accredited ethical committee within 15 days, including the reasons for the premature termination.

Within one year after the end of the study, the responsible researcher will submit a final study report with the results of the study, including any publications/abstracts of the study, to the accredited ethical committee.

Public disclosure and publication policy:

Public disclosure and publication policy is regulated by InSup-C. Dissemination Strategy (October 2013), available at request. An outline publication timeline with suggested topics, lead work package author and scientific target journals is detailed in the Dissemination Strategy. An interactive website has been developed. The website will signpost study results as these become available.

Monitoring level related to risk classification:

As in the previous section it was estimated that this study has a negligible risk, minimal monitoring will take place. Table 4 displays the activities the monitor will perform. Monitoring will be conducted by a qualified monitor who has knowledge of current legislation and regulation and who is independent from this study. Findings will be reported to the coordinating investigator of the Radboud umc in a fixed format. If the monitor identifies substantial and/or frequent faults, this will be reported to the head of the department and/or the company board.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 year or above
2. Able to communicate in the national language (Dutch, English, German, Hungarian)
3. Cognitively able to complete questionnaires and to participate in interviews.

   Additional inclusion criteria for patients:
4. Surprise question "Would the patient's attending doctor be surprised if the patient died within 1 year?" is answered "No" by the patient's attending doctor
5. Patients need to meet on of the following clinical criteria:

   * Malignant disease: Advanced cancer (cancer with local progression and / or distant metastasis at presentation).
   * Chronic Heart Failure: Severe heart failure (in accordance with New York Heart Association (NYHA) classification stage III-IV)
   * COPD: Gold stage IV classification

Exclusion criteria:

1. People who lack mental capacity to give interviews and fill in questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In Belgium, Germany, Hungary, The Netherlands and United Kingdom 3-5 'model initiatives' of palliative care were selected. From each initiative, patients with advanced cancer, COPD and CHF, their family and professional caregivers are recruited. Patients (and if presented the family caregiver) are recruited by their main responsible doctor or (research) nurse involved in the initiative under examination. Participants need to meet the inclusion and exclusion criteria in order to be eligible for the study. A family caregiver is defined as the person who takes care and supports the patient for most of the time. Family caregivers are not necessarily a family member. Professional caregivers involved in the IPC initiatives under examination are invited for the group interviews.
Sampling Method: Non-Probability Sample
Enrollment: 576 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Experiences with IPC initiatives at 3 months | Baseline and Month 3
  The semi-structured interviews will be used to explore views of patients and family caregivers about their experiences with the integrated palliative care initiative. Topics include:
  * An exploration of problems and needs of the patient
  * An exploration of the contacts and relationships of patients and family caregivers with professional caregivers
  * An exploration of satisfaction and perceived deficits in service provision from the perspective of patients and family caregivers
  * An exploration of the views of patients and family caregivers on collaboration between professional care providers in the care network of the patient.
Change from baseline Quality of care at 1, 2 and 3 months | Baseline, Month 1, Month 2, Month 3
  Quality of care/satisfaction will be measured using the Canhelp Lite and the Social Network Analysis (SNA) method.
  Outcomes will be explored in the interviews, see also "Experiences with IPC initiatives"
Change from baseline Quality of life at 1, 2, and 3 months | Baseline, Month 1, Month 2, Month 3
  Quality of Life will be measured using the Palliative Care Outcome Scale (POS) version 1.
  Outcomes will be explored in the interviews, see also "Experiences with IPC initiatives"
Change from baseline Perceived symptoms at 1, 2, and 3 months | Baseline, Month 1, Month 2, Month 3
  Quality of Life will be measured using the Palliative Care Outcome Scale (POS) version 1.
  Outcomes will be explored in the interviews, see also "Experiences with IPC initiatives".
Change from Perceived collaboration between professional caregivers at 3 months | Baseline, Month 3
  Quality of Life will be measured using Social Network Analysis method (SNA). Outcomes will be explored in the interviews, see also "Experiences with IPC initiatives"
Change from baseline Burden and rewards of care giving at 1, 2, and 3 months | Baseline, Month 1, Month 2, Month 3
  Burden and rewards of care giving will be measured using the Caregiver Reaction Assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Marieke Groot, PhD, Principal Investigator — Radboud University Medical Center
Locations (5):
- Katholieke Universiteit Leuven, Leuven, Belgium
- University Hospital Bonn, Bonn, Germany
- Medical University of Pecs, Pécs, Hungary
- Radboud University Medical Centre Palliative consultation team, Nijmegen, Gelderland, Netherlands
- Lancaster General Hospital, Lancaster, United Kingdom